CLINICAL TRIAL: NCT00264407
Title: Age-Related Hearing Loss: Presbycusis & Its Neural Bases
Brief Title: Neural Changes in the Aging Auditory System
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: Rochester Institute of Technology (Other); National Institute on Aging (NIA) (NIH); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Other Study IDs: 10121; P01AG009524 (NIH)
Record Dates: First submitted 2005-12-08; First posted 2005-12-12 (Estimated); Last update posted 2005-12-12 (Estimated); Status verified 2005-12

CONDITIONS: Progesterone; Estrogens; Hearing; Psychoacoustics; Auditory Perceptual Disorders
Keywords: Hearing Loss, Central; Presbycusis; Hearing Loss, Sensorineural; Hearing Loss, Cochlear; Hearing Loss, Bilateral; Sex Steroid Hormones; Estradiol
MeSH Terms: conditions — Auditory Perceptual Disorders; Hearing Loss, Central; Presbycusis; Hearing Loss, Sensorineural; Hearing Loss, Bilateral | interventions — Hormone Replacement Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

INTERVENTIONS:
Drug: Hormone Replacement Therapy - HRT

SUMMARY:
The purpose of this study was to determine the effects of hormone replacement therapy (HRT) on hearing in post-menopausal women.

DETAILED DESCRIPTION:
Background: Female hormone influences on the development and aging of the auditory system are not completely understood. The present study retrospectively analyzed and compared hearing abilities among post-menopausal women taking hormone replacement therapy (HRT), treated with estrogen and progesterone (E+P); estrogen alone (E), and a third (control - NHRT) group, matched for age, who did not receive any HRT.

Methods: 126 subjects, (60-86 yr), N=32, E+P; N=31, E; N= 63, NHRT; matched for age and health status participated. All had relatively healthy medical histories, absence of significant noise exposure, middle ear problems, major surgeries or current/heavy smoking. Hearing tests included pure tone audiometry (PTA), tympanometry, distortion-product otoacoustic emissions (DPOAEs), transient otoacoustic emissions (TEOAEs) and hearing-in-noise-test (HINT). The latter is a test for speech perception in background noise: the major complaint of hearing-impaired persons.

.

ELIGIBILITY:
Inclusion Criteria:

* Healthy middle ears

Exclusion Criteria:

* ototoxic medications
* serious medical health problems
* neurological conditions
* Meniere's disease or labyrinthitis
* those who failed cognitive screening tests (Mini-Mental Test)
* current/heavy smokers
* conductive hearing loss
* history of noise damage and/or audiograms signifying noise damage
* poor speech discrimination scores (80% or less)

Ages: 60 Years to 86 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126
Dates: Start 2001-01; Study Completion 2005-02

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Frisina, Ph.D., Study Director — University of Rochester Medical School
Locations (2):
- United States (2):
  - International Center Hearing & Speech Research - NTID - RIT, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York